CLINICAL TRIAL: NCT06488196
Title: Feasibility, Acceptability, and Fidelity of Motivational Interviewing Targeting Ethnically-, Linguistically-, and Racially-diverse Mothers' Neonatal Intensive Care Unit (NICU) Bedside Presence
Brief Title: Feasibility, Acceptability, and Fidelity of Motivational Interviewing to Increase Maternal NICU Presence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00182045
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Neonatal Intensive Care
Keywords: motivational interviewing; NICU
MeSH Terms: interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Intervention Model Description: The investigators used a randomized controlled trial (RCT) design and randomized consenting mothers (1:1) in blocks of 10 to the MI-arm or a treatment-as-usual (TAU) control-arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Mothers in the MI-arm received up to six weekly MI sessions until the baby was discharged from the NICU. Mothers whose baby was discharged prior to or during week six completed measures at enrollment and NICU discharge. Mothers whose baby was discharged after week six completed questionnaires at enrollment and at the end of week six. Mothers could choose whether to complete MI in English or Spanish. Native Spanish-speaking, ethnically-matched providers conducted Spanish-language sessions. Study team members offered to read questionnaires aloud and record responses; however, all participants chose to independently complete paper-and-pencil measures.
  Interventions: Behavioral: Motivational Interviewing
- Treatment as Usual (Active Comparator): In the institution in which the investigators conducted this study, per institutional standards, TAU included the opportunity for mothers to meet with a NICU psychologist or psychology trainee at least once-per-week for supportive care.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational interviewing (MI) is a person-centered, goal-oriented psychotherapeutic intervention designed to enhance the recipient's motivation for and commitment to a target behavior or behavior change. MI's core action mechanisms include strengthening the recipient's change talk (e.g., assertions about desire and commitment toward the target behavior) and softening the recipient's sustain talk (e.g., statements about barriers). MI clinicians achieve these goals using specific micro-skills (e.g., reflective listening) that reflect MI's fundamental spirits (i.e. collaboration, acceptance, compassion, evocation.
  Arms: Motivational Interviewing
Other: Treatment As Usual — TAU included the opportunity for mothers to meet with a NICU psychologist or psychology trainee at least once-per-week for supportive care.
  Arms: Treatment as Usual

SUMMARY:
Maternal presence in the NICU during an infant's hospitalization is critical for the infant's medical recovery and overall neurodevelopmental trajectory. However, despite the importance of maternal presence in these settings, the current literature shows that families are often absent at bedside. To date, no behavioral interventions have been conducted to promote increased maternal visitation patterns in NICU settings. This project will aim to fill this gap in the literature by conducting a pilot study that uses a motivational interviewing intervention with the aim of increasing maternal visitation rates to a level IV NICU.

DETAILED DESCRIPTION:
This study will be conducted as a randomized controlled pilot trial of a motivational interviewing intervention. Mothers will be contacted for enrollment in the study within the first 48-72 hours of the infant's NICU admission. Contact with the mother will occur in-person within those first 48-72 hours of admission. If mother is unavailable in person within the first 72 hours, a telephone call will be made to her. Should the mother agree to participate in the study, written consent will be obtained if the meeting is taking place in person. If the first contact takes place via telephone, then verbal consent alone will be obtained at that time followed by written consent during the first in-person meeting with mother (see below for detailed consent procedures). Once enrolled, the mother will be assigned to one of two study arms - the treatment group or the treatment-as-usual (comparison) group. Mothers will not be provided with information about study arm assignment.

Cluster randomization: Group assignment will be determined by location of the infant in the NICU. The comparison group will be assigned to the North side of the unit while the treatment group will be assigned to the South side of the unit. Assignment to each side of the unit (i.e., North or South) is routinely determined based on census capacity/availability and not based on other factors that may inhibit the randomization process.

Both study groups will receive 6 sessions with the experimental group receiving motivation interviewing (MI) and the control group receiving support as usual. Additional supportive interventions will continue as needed and determined by the clinical needs and consistent with current treatment as usual (TAU). All families will also complete a discharge study visit within 7 days of NICU discharge; hence, participants will receive a total of at least 7 study visits throughout infant's hospitalization. The goal of the first session will be to establish rapport and obtain information about the sources of stress and distress to target in later sessions. Weekly follow-up visits with all families will continue utilization of supportive and problem-solving approaches to manage stressors identified in the initial session. If mothers cannot be reached in person for projected visits at various time points, attempts will be made to connect with mothers via telephone irrespective of study assignment.

More specifically, the first consultation will consist of a semi-structured clinical interview that will assess the following general topics: (1) family-reported psychosocial factors related to the perinatal period (i.e., antepartum, labor/delivery, postpartum, NICU hospitalization, possible NICU discharge periods); (2) perceptions of the caregiver-infant relationship; (3) family psychosocial stressors; (4) family adjustment to the NICU setting; (5) family self-report of coping; (6) family self-report of barriers to visiting the NICU.

All sessions will be audio-recorded in the treatment arm of the study while a portion of the sessions will be recorded in the comparison group (see data analysis section). All audiotaped sessions will be reviewed for fidelity to motivational interviewing treatment protocol by an MI-certified trainer for English sessions while the Spanish sessions will be reviewed by a doctoral-level graduate student with training in MI and under the supervision of the certified trainer reviewer.

However, if mother does not finish the questionnaires by the end of the visit/contact, she may be asked to stay longer at the unit or on the phone to complete the remaining questions. If she does not have time to complete the questions, the investigators will develop a plan for completing the remaining questions. For instance, the investigators may ask to contact her via phone within the next five days in order to read and complete the remaining questions or meet again during the next visit to the NICU.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking mothers >18 years-old with a NICU-hospitalized infant

Exclusion Criteria:

* Suicidality, cognitive disability preclude consent/participation, or psychotic/manic symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers of infants hospitalized in the NICU
Enrollment: 95 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Feasibility, as assessed by >75% of MI-randomized mothers receiving at least one MI session | 3 years
  Feasibility as assessed by >75% of MI-randomized mothers receiving > one MI session

SECONDARY OUTCOMES:
Acceptability as assessed by the number of mothers' open to completing additional MI session/s | 3 years
  MI acceptable, as evidenced by mothers reporting willingness (yes/no) to receive a second MI session after completing their first MI session.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Faith, PhD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No